CLINICAL TRIAL: NCT02671240
Title: Prognosis of Behavioral Addiction in Parkinson's Disease
Acronym: PROBA-PD
Status: Terminated | Type: Observational
Why Stopped: Investigator's decision
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6246
Record Dates: First submitted 2016-01-18; First posted 2016-02-02 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Addiction
Keywords: Parkinson disease; behavioral addiction; akinéto-rigid syndrome; dopamine agonist
MeSH Terms: conditions — Behavior, Addictive; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- - Patients with behavioral addiction
- - Patients with no behavioral addiction

SUMMARY:
Our hypothesis is that the conventional treatment of Behavioral Addiction in Parkinson's disease is often not effective, and that affects the motor aspects (worsening akinéto-rigid syndrome and / or worsening of dyskinesia due to higher levodopa doses to compensate for the drop in behavioral addictions) and non-motor (withdrawal syndrome dopamine agonist) anxiously including apathy.

Our goal is to describe the natural history of Behavioral Addiction under the effect of the evolution of the disease and adapt treatment according to the prior art, through a study of a larger population of patients than in the few published studies.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 30 years
* Parkinson's disease according to the criteria of UKPDSBB
* Time evolution of the top disease or equal to 5 years

Exclusion criteria:

* Lack of Parkinson's disease and atypical parkinsonism
* Patient not previously included in PD-BADGE

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease who developed or not a behavioral addiction
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Survival time before disappearance of behavioral addiction defined by a score of less than 2 on the scale of behavioral assessment of Parkinson's disease | 12 months after selection

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ANHEIM, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Neurologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No